CLINICAL TRIAL: NCT05874726
Title: Biological Sample Repository for Gastrointestinal Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Pichamol Jirapinyo, MD, MPH (Other)
Collaborators: Tufts University (Other); Boston Children's Hospital (Other); Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Pichamol Jirapinyo, MD, MPH, Associate Director of Bariatric Endoscopy, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Other Study IDs: 2022P003060
Record Dates: First submitted 2023-03-31; First posted 2023-05-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Obesity, Morbid; Obesity, Primary; Gastro-Intestinal Disorder; Overweight and Obesity; Overweight; Overweight or Obesity; Diabetes Type 2; Diabetes Mellitus; Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias; Sleep Apnea; GERD; Gastroesophageal Reflux; Musculoskeletal Pain Disorder; Cancer
Keywords: Gut Hormones; Bariatric Surgery; Weight Loss; Weight Loss Diets; Anti-obesity Medications; Endoscopic Metabolic and Bariatric Therapies (EMBT); Bariatric Endoscopy; Intragastric balloon (IGB); Ablation Techniques; Submucosal Tunneling Procedures; pylorus sparing antral myotomy (PSAM); gastroplasty with endoscopic myotomy (GEM); Gastric peroral endoscopic myotomy (G-POEM); Tissue Plication; Primary Obesity Surgery Endolumenal (POSE); Restorative Obesity Surgery Endoluminal (ROSE); Endoluminal sleeves; Endoscopic Suturing; Endoscopic Sleeve Gastroplasty (ESG); laparoscopic adjustable gastric banding (LAGB); laparoscopic sleeve gastrectomy (LSG); Roux-en-Y gastric bypass (RYGB); bilio-pancreatic diversion (BPD); bilio-pancreatic diversion with duodenal switch (BPD-DS); Pathophysiology of obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid; Digestive System Diseases; Overweight; Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension; Hyperlipidemias; Sleep Apnea Syndromes; Gastroesophageal Reflux; Collagen Diseases; Neoplasms; Weight Loss | interventions — Blood Specimen Collection; Urine Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — * Blood (serum will be extracted and stored at -80⁰C),
  * Urine (stored at -80⁰C),
  * Tissue (gastric, duodenum, jejunum and ileum - number of biopsies will be 3-4 from each site, ranging in size from 4-7mm) - These samples collected will be extra biopsies that are taken for research purposes during a clinically planned endoscopy for which biopsies are being planned.
  * Data from medical records will be collected including: age, gender, vitals, weight, bmi, graphs, medical history, surgical history, endoscopy reports, radiology reports, labs, demographics, medications, problem list. Investigators do plan to continue collecting data into the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bariatric Surgery Patients: Subjects who have had bariatric surgery for obesity - primary and revision. Bariatric surgical procedures include laparoscopic adjustable gastric banding (LAGB), laparoscopic sleeve gastrectomy (LSG), Roux-en-Y gastric bypass (RYGB), bilio-pancreatic diversion (BPD) with or without duodenal switch (BPD-DS).
  Interventions: Diagnostic Test: Blood Collection; Diagnostic Test: Urine Collection; Diagnostic Test: Tissue Sample Collection
- Endoscopic Metabolic and Bariatric Therapies: Subjects who have had endoscopic bariatric therapies for obesity - primary and revision. Bariatric endoscopic procedures include ablation techniques, intragastric balloons, submucosal tunneling procedures (PSAM, GEM, G-POEM), tissue plication platforms (POSE, ROSE), endoluminal sleeves and endoscopic suturing devices (ESG).
  Interventions: Diagnostic Test: Blood Collection; Diagnostic Test: Urine Collection; Diagnostic Test: Tissue Sample Collection
- Medical Management: Subjects who follow lifestyle modification and/or anti-obesity medications for treatment of obesity with no previous surgical intervention for obesity. Medical therapies include weight loss diets or anti-obesity medications.
  Interventions: Diagnostic Test: Blood Collection; Diagnostic Test: Urine Collection; Diagnostic Test: Tissue Sample Collection

INTERVENTIONS:
Diagnostic Test: Blood Collection — Blood collection via venipuncture
Diagnostic Test: Urine Collection — Free catch urine sample collection
Diagnostic Test: Tissue Sample Collection — Tissue (gastric, duodenum, jejunum and ileum - number of biopsies will be 3-4 from each site, ranging in size from 4-7mm) - These samples collected will be extra biopsies that are taken for research purposes during a clinically planned endoscopy for which biopsies are being planned.
  Other Names: Biopsy

SUMMARY:
The goal of this observational study has the purpose of collecting biological samples from obese patients undergoing evaluation for weight loss by means of medical or endoscopic therapies; and of post bariatric surgery patients presenting with short- and long-term surgical complications. The aim is to enhance the overall understanding of the mechanisms leading to obesity, weight loss, failure to lose weight, and weight regain following treatment. Additional goals are to determine the efficacy of endoscopic and surgical procedures, to identify potential therapeutic targets and disease biomarkers that predict response to therapy.

DETAILED DESCRIPTION:
The prevalence of obesity in the U.S. has reached unacceptably high numbers over the past three decades. Approximately 68% of the American population over the age of 20 is overweight, while 35.7% meet criteria for obesity (CDC). Obesity has become a leading cause of morbidity, mortality and reduced quality of life; and places patients at high risk for several chronic conditions, including: diabetes (DM), hypertension (HTN), hyperlipidemia (HL), sleep apnea, GERD, musculoskeletal disorders and cancer. In addition, obesity imposes a major burden in the American healthcare system, with an estimated annual cost of 147 billion U.S. dollars.

Treatment of obesity is challenging. Preventive measures and medical therapy have not been effective in fighting this epidemic. Diet and exercise, though logical, are hindered by high recidivism and a propensity to regain weight to pre-weight loss levels. Anti-obesity drugs are largely ineffective and limited by safety and side-effects profile. Even bariatric surgery, which provides significant and rapid weight loss, is still followed by substantial weight regain over time. In addition, surgery is associated with a 1% mortality risk, 5-25% 1-year morbidity, and is not readily accessible. Fewer than 1% of eligible obese patients undergo surgery each year. In face of all these challenges, there is an urgent need to better understand the pathophysiology of obesity and the effects of current weight loss interventions. This knowledge will provide a new framework for the development of more effective preventive measures and therapies.

The pathophysiology of obesity is complex. Weight gain results from an energy imbalance; that is, when energy intake is higher than expenditure. In this context, obesity has been attributed to a shift in diet toward increased consumption of energy-dense foods, and to sedentary lifestyle. However, little is known about the physiological mechanisms underlying this trend, which are thought to be regulated by genetic, metabolic and neurobehavioral factors. Even less is understood on how increased adiposity leads to the development of many metabolic disorders, including DM. Surprisingly, these mechanisms can be reversed by bariatric procedures, which in addition to weight loss, have dramatic beneficial effects on metabolic disorders such as DM, HTN, and HL. Therefore, surgery has become an important study tool to enhance our understanding of the pathophysiology of obesity. The collection of biological samples from patients before and after weight loss therapies, including endoscopic and surgical procedures, will provide the basis for a series of studies that will focus on investigating:

* the mechanisms that lead to obesity, particularly appetite and gut regulatory peptides;
* the clinical, physiological, hormonal and metabolic changes imposed by medical, surgical and endoscopic procedures to treat obesity;
* the mechanisms of weight regain following bariatric surgery;
* the mechanism of failure to lose weight following endoscopic or surgical procedures;
* the effects of endoscopic procedures on weight regain following bariatric surgery;
* biomarkers that predict response to medical, endoscopic and surgical therapies;
* biomarkers that predict weight regain or therapeutic failures;
* novel therapeutic targets for the treatment of obesity.

Medical therapies include weight loss diets or anti-obesity medications. Bariatric endoscopic procedures include ablation techniques, intragastric balloons, submucosal tunneling procedures (PSAM, GEM, G-POEM), tissue plication platforms (POSE, ROSE), endoluminal sleeves and endoscopic suturing devices (ESG).

Bariatric surgical procedures include laparoscopic adjustable gastric banding (LAGB), laparoscopic sleeve gastrectomy (LSG), Roux-en-Y gastric bypass (RYGB), bilio-pancreatic diversion (BPD) with or without duodenal switch (BPD-DS).

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years of age,
* Suffer from obesity, defined by BMI≥30 kg/m2 (body mass index: weight in kilograms divided by the square of the height in meters).

Exclusion Criteria:

* Positive laboratory tests for any of the following pathogens: Hepatitis B virus (HBV); Hepatitis C virus (HCV); Human Immunodeficiency Virus Types 1 and 2 (HIV); Human T-Lymphotropic virus Types I and II (HTLV); Treponema pallidum (syphilis); Clostridium Difficile (C. Diff)
* History of gastrointestinal malabsorptive disorders including a known history of celiac disease, and/or chronic pancreatitis,
* History of any inflammatory disease of the gastrointestinal tract,
* Patient is of childbearing age and not practicing effective birth control method, pregnant or lactating
* History of a myocardial infarction or cerebro-vascular accident in the last year, or history of unstable cardiovascular disease,
* History of cancer or life expectancy of < 2 yrs,
* Use of any medications (prescription or OTC), including herbal or other supplements for treatment of obesity,
* History of known hormonal or genetic cause for obesity,
* History of any psychiatric disorders including dementia, active psychosis, severe depression requiring > 2 medications, history of suicide attempts, alcohol or drug abuse within the previous 12 months,
* Any condition or major illness that, in the investigator's judgment, places the subject at undue risk of participating in the repository,
* Unable to understand the risks, realistic benefits and requirements of the repository,
* Use of investigational therapy or participation in any other clinical trial within 12 weeks prior to signing the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this repository is to study obesity, as well as the effects of weight loss therapies on several clinical, physiological, hormonal and biochemical parameters. Therefore, enrollment in this repository will be limited to patients with obesity undergoing evaluation for weight loss through medical, endoscopic or surgical means. Obesity is a condition that affects all ethnic and racial groups. Investigators do not anticipate that any particular group of patients will be disproportionately represented. Although obesity affects both children and adults, this repository will be limited to adult patients, which represent the practices of the physicians involved in this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Serum sample repository | Change from Baseline to 10 years.
  Blood (10 ml) will be collected from the enrolled subjects, serum will be extracted and stored at -80 degrees for up to 10 years.
Urine sample repository | Change from Baseline to 10 years.
  Urine (5 ml) will be collected via free catch method and stored at -80 degrees C for up to 10 years.
Tissue sample repository | Change from Baseline to 10 years.
  Tissue samples (gastric, duodenum, jejunum and ileum - number of biopsies will be 3-4 from each site, ranging in size from 4-7mm) will be collected during a scheduled endoscopic examination. Biopsy tissue will be collected with a large capacity biopsy forceps and deposited into a conical vial containing a freshly prepared balanced salt solution including a HEPES buffer at the bedside, using 5mL of buffered salt solution per 5-10 mm3 of tissue biopsy, at 4 degrees C. Tissue will be stored at -80⁰C until they are "used up" or for up to 10 years from collection.

CONTACTS AND LOCATIONS:
Overall Officials: Pichamol Jirapinyo, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
MGB and non-MGB investigators may request samples (any of the samples listed in this protocol) from this tissue repository. This request will be made after establishing a formal collaboration with investigators in this protocol. Requests will be made in the form of a written document stating the title and purpose of the project, as well as which experimental procedures will be done with the repository samples. In addition to a written request, collaborators will have to share their approved IRB protocol with the investigators in this repository.
Supporting Information: Study Protocol
Time Frame: 12 months after publication
Access Criteria: Requests will be overseen by Michele Ryan, the research coordinator and laboratory manager. Requests will be reviewed by the PI, and approved based on her judgment and the lack of conflicts with the PI's current research studies.
  Michele Ryan and Dr. Jirapinyo will assess all tissue requests and ensure a current, IRB-approved protocol is in place covering the proposed research.
  For non-MGB investigators that are not part of the study team, tissue will only be distributed that is coded, but not directly identifiable. Investigators will not allow the recipient researcher to identify the individual from whom the tissue was obtained. Investigators will have the recipient researcher agree in writing never to attempt to access identifiable health/medical information or to attempt to identify and contact the individual(s) who have provided the samples.

REFERENCES:
- [Background] Ogden CL, Yanovski SZ, Carroll MD, Flegal KM. The epidemiology of obesity. Gastroenterology. 2007 May;132(6):2087-102. doi: 10.1053/j.gastro.2007.03.052. PMID 17498505
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Powell AG, Apovian CM, Aronne LJ. New drug targets for the treatment of obesity. Clin Pharmacol Ther. 2011 Jul;90(1):40-51. doi: 10.1038/clpt.2011.82. Epub 2011 Jun 8. PMID 21654742
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Dixon JB, Lambert GW. The obesity paradox--a reality that requires explanation and clinical interpretation. Atherosclerosis. 2013 Jan;226(1):47-8. doi: 10.1016/j.atherosclerosis.2012.11.005. Epub 2012 Nov 15. No abstract available. PMID 23219371
- [Background] Guyenet SJ, Schwartz MW. Clinical review: Regulation of food intake, energy balance, and body fat mass: implications for the pathogenesis and treatment of obesity. J Clin Endocrinol Metab. 2012 Mar;97(3):745-55. doi: 10.1210/jc.2011-2525. Epub 2012 Jan 11. PMID 22238401
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery Worldwide 2008. Obes Surg. 2009 Dec;19(12):1605-11. doi: 10.1007/s11695-009-0014-5. PMID 19885707
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Perdomo CM, Cohen RV, Sumithran P, Clement K, Fruhbeck G. Contemporary medical, device, and surgical therapies for obesity in adults. Lancet. 2023 Apr 1;401(10382):1116-1130. doi: 10.1016/S0140-6736(22)02403-5. Epub 2023 Feb 9. PMID 36774932
- [Background] Qureshi H, Saeed N, Jovani M. Updates in Endoscopic Bariatric and Metabolic Therapies. J Clin Med. 2023 Jan 31;12(3):1126. doi: 10.3390/jcm12031126. PMID 36769774
- [Background] Jirapinyo P, Thompson CC. Primary Bariatric Procedures. Dig Dis Sci. 2022 May;67(5):1674-1687. doi: 10.1007/s10620-022-07393-z. Epub 2022 Mar 29. PMID 35348970
- [Background] Dolan RD, Schulman AR. Endoscopic Approaches to Obesity Management. Annu Rev Med. 2022 Jan 27;73:423-438. doi: 10.1146/annurev-med-042320-125832. Epub 2021 Sep 23. PMID 34554827